CLINICAL TRIAL: NCT03955198
Title: A Multicentric Phase II Trial of Stereotactic Radiotherapy Plus Durvalumab Continuation for Patients With NSCLC Metachronous Oligometastatic Disease Under Durvalumab Consolidation Following Chemoradiation
Brief Title: A Trial Evaluating Stereotactic Radiotherapy Plus Durvalumab Continuation for Patients With NSCLC Metachronous Oligometastatic Disease Under Durvalumab Consolidation Following Chemoradiation
Acronym: SILK BM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18POUM06
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: NSCLC
Keywords: NSCLC; Anti-PD-L1; Durvalumab; Stereotactic Radiation therapy; Oligometastatic disease
MeSH Terms: interventions — Radiotherapy; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with NSCLC metachronous oligometastatic disease (Experimental)
  Interventions: Combination Product: Radiotherapy + durvalumab

INTERVENTIONS:
Combination Product: Radiotherapy + durvalumab — Radiotherapy will be administered in combination with Durvalumab

SUMMARY:
This study is a single-arm phase II, multicenter study designed to evaluate the activity of stereotactic radiotherapy plus the continuation of durvalumab for 12 more months for patients presenting with NSCLC metachronous oligometastatic disease during post-chemoradiotherapy durvalumab consolidation.

Fifty patients will have to be enrolled in this phase II trial.

Total duration of treatment will be 12 months.

Patients will be followed for a maximum of 2 years following the date of inclusion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
2. Under durvalumab consolidation following chemoradiotherapy (sequential or concurrent) for previous stage III NSCLC ; patients must have received at least one infusion of durvaluamb consolidation and should be within 12 months of the first infusion ; the last infusion should have been performed within the last 28 days
3. While receiving durvalumab, patients must not have experienced ≥Grade 3 immune related adverse event. Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic. Patients must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE
4. No history of previous metastatic disease
5. Stage IV metastatic disease
6. Patients with 1 to 5 metastases in total, in no more than 3 organs (including brain) documented on the basis of contrast-enhanced CT-scanner of the chest, abdomen and pelvis, 18FDG-PET and brain MRI (and liver MRI in case of liver metastases)
7. All metastatic lesions are less of 4 cm in greater diameter
8. For patients with brain metastases : surgery of one or several brain lesion(s) is allowed before enrollment provided that there is at least one associated non-resected lesion (cranial or extra-cranial)
9. All lesions are amenable to SRT in terms of dose constraints to the organs at risk, with no prior radiotherapy interfering with SRT
10. No local relapse (in-field) or regional mediastinal relapses associated
11. Patient with wild type EGFR and ALK
12. Age ≥ 18 years at time of study entry
13. ECOG performance status < 2 i.e. 0 or 1
14. Body weight >30kg
15. Life expectancy of at least 3 months
16. Adequate Hematology laboratory data within 6 weeks prior to start of treatment: Absolute neutrophils> 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hemoglobin ≥ 9 g/dL
17. Adequate Biochemistry laboratory data within 6 weeks prior to start of treatment: Total bilirubin ≤ 1.5 x ULN (except patient with confirmed Gilbert's syndrome or liver metastasis: Total bilirubin ≤ 3 X ULN), Transaminases ≤ 2.5 x ULN, Alkalin phosphatases ≤ 5 x ULN, Creatinine clearance > 40 mL/min (Cockcroft)
18. Women should be post-menopaused or willing to accept the use an effective contraceptive regimen during the treatment period and at least 3 months after the end of the study treatment. All non-menopaused women should have a negative pregnancy test within 72 hours prior to registration. Men should accept to use an effective contraception during treatment period and at least 3 months after the end of the study treatment
19. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
20. Signed written informed consent
21. Patient affiliated to a Social Health Insurance in France

Exclusion Criteria:

1. Cancer histology other than NSCLC
2. Local relapse or mediastinal relapse associated to oligometastatic relapse following chemoradiation
3. Prior radiotherapy near the metastatic lesions precluding ablative SRT
4. Contraindication to SRT of a lesion due to organ dysfunction; in particular, patients with lung lesions and documented or suspected interstitial lung disease should not be included
5. Metastatic spinal cord compression
6. Brain metastases in the brainstem
7. Known leptomeningeal metastases
8. Patient unable to have MRI for any reason (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity)
9. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician
10. Participation in another therapeutic trial within the 30 days prior to entering this study (participation in a survival follow-up period of a clinical study is not an exclusion criterion)
11. Prior therapy with an anti-PD-1, anti-PD-L1 (except during durvalumab consolidation), anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
12. Current or prior use of immunosuppressive medication within 7 days before the first fraction of RT; however the use of corticosteroids at any dose for the management of an AE or a compressive progressive lesion is allowed
13. Active suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, diverticulitis with the exception of diverticulosis, systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). Note: participants with vitiligo or alopecia, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, patients with celiac disease controlled by diet alone, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger, are permitted to enroll
14. Known primary immunodeficiency or active HIV (positive HIV 1/2 antibodies)
15. Known active or chronic viral hepatitis or history of any type of hepatitis within the last 6 months indicated by positive test for hepatitis B surface antigen (HBV sAG) or hepatitis C virus ribonucleic acid (HCV antibody)
16. History of active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
17. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
18. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
19. History of severe allergic reactions to any unknown allergens or any components of the study drug
20. History of allogenic organ transplantation
21. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP
22. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab
23. Patient who has forfeited his/her freedom or who is under legal protection (curatorship and guardianship, protection of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Progression-free survival defined as the time from inclusion to disease progression (per RECIST v1.1) or death from any cause, whichever occurs first. | 24 months for each patient

SECONDARY OUTCOMES:
Immune progression-free survival defined as the time from inclusion to disease progression (per iRECIST) or death from any cause, whichever occurs first. | 24 months for each patient
Safety will be assessed by the toxicity grading of the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v 5.0). | 24 months for each patient
Quality of life will be evaluated using the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30). | 24 months for each patient

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Institut de Cancérologie de Bourgogne - Auxerre, Auxerre
  - Institut Sainte-Catherine, Avignon
  - Centre François Baclesse, Caen
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Hospitalier Universitaire Lyon Sud, Lyon
  - Centre Henri Becquerel, Rouen
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse